CLINICAL TRIAL: NCT01508650
Title: Rehabilitation and Exercise Training After Hospitalization: Assessing Benefit in Acute Heart Failure (REHAB-HF) Pilot Study
Brief Title: Rehabilitation and Exercise Training After Hospitalization
Acronym: REHAB-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00016973
Record Dates: First submitted 2011-12-21; First posted 2012-01-12 (Estimated); Results first posted 2019-02-07 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2018-09

CONDITIONS: Heart Failure
Keywords: heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No intervention (Active Comparator): Usual care control group
  Interventions: Behavioral: Usual care
- Active Comparator (Active Comparator): Multi domain rehabilitation intervention
  Interventions: Behavioral: Rehabilitation intervention

INTERVENTIONS:
Behavioral: Usual care — Usual care control group
  Arms: No intervention
Behavioral: Rehabilitation intervention — Multi-domain rehabilitation intervention
  Arms: Active Comparator

SUMMARY:
Rehabilitation and Exercise Training after Hospitalization: Assessing Benefit in Acute Heart Failure (REHAB-HF) pilot is a multi-site, randomized clinical pilot study designed to establish the feasibility of conducting a larger clinical trial to address the hypothesis that, in addition to standard care, a novel, progressive, multi-domain 3-month rehabilitation intervention administered to elderly patients with acute decompensated heart failure (ADHF) will improve key clinical outcomes, including the rate of rehospitalization and death, physical function, and quality of life.

DETAILED DESCRIPTION:
Three centers,Wake Forest Baptist Health along with Thomas Jefferson University Hospital-Co-Investigator Dr. David Whellan, and Duke Medical Center- Co-Investigator Dr. Christopher O'Connor, will recruit a total of 60 consenting patients ≥ 60 years old hospitalized with ADHF. Once identified and screened, the participants will be randomized in a 1:1 fashion to receive a 3 month novel rehabilitation and exercise training intervention or usual care. This multi-domain intervention will include endurance, mobility, strength, and balance training and be tailored based on participant performance in each of these domains. It will begin during the hospitalization and continue three times per week in an outpatient facility.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years old
* Hospitalized for the management of ADHF or diagnosed with ADHF after being hospitalized for another reason. ADHF will be defined as a combination of symptoms, signs, and HF-specific medical treatments.

Exclusion Criteria:

* Planned discharge other than to home or a facility where the participant will live independently.
* Acute myocardial infarction
* Already participating in cardiac rehabilitation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-10; Primary Completion 2012-06-08 (Actual); Study Completion 2012-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dalane W Kitzman, MD, Principal Investigator — Wake Forest Baptist Hospital
Locations (3):
- United States (3):
  - Duke Medical Center, Durham, North Carolina
  - Wake Forest Baptist Hospital, Winston-Salem, North Carolina
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Reeves GR, Whellan DJ, O'Connor CM, Duncan P, Eggebeen JD, Morgan TM, Hewston LA, Pastva A, Patel MJ, Kitzman DW. A Novel Rehabilitation Intervention for Older Patients With Acute Decompensated Heart Failure: The REHAB-HF Pilot Study. JACC Heart Fail. 2017 May;5(5):359-366. doi: 10.1016/j.jchf.2016.12.019. Epub 2017 Mar 8. PMID 28285121

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Intervention | Active Comparator
Started | 12 | 15
Completed | 12 | 12
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Intervention | Active Comparator | Total
Number analyzed (Participants) | 12 | 15 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.8 (10.8) | 72.7 (9.1) | 72.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 4 | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 15 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 8 | 15
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 6 Minute Walk Test
Description: The 6 minute walk test submaximal exercise test that measures how far a participant can walk in 6 continuous minutes. Participants are instructed to walk as far as possible in 6 minutes, and are allowed to slow down and take breaks as needed due to symptoms.
Time Frame: up to 3 months
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | No Intervention | Active Comparator
Number analyzed (Participants) | 12 | 12
meters | 224 (22) | 247 (22)

2. Secondary Outcome: SPPB (Short Physical Performance Battery)
Description: The SPPB is a multi-component measure of physical function. The SPPB is composed of 3 components-standing balance, gait speed, and timed repeated chair rise-each scored on a scale from 0 to 4 and combined for a total score of 0 to 12. A higher score denotes better physical function.
Time Frame: up to 3 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | No Intervention | Active Comparator
Number analyzed (Participants) | 12 | 12
units on a scale | 6.3 (0.5) | 7.4 (0.5)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | No Intervention | Active Comparator
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/15
Serious Adverse Events (participants affected / at risk) | 8/12 | 11/15
Other Adverse Events (participants affected / at risk) | 2/12 | 5/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Intervention (N=12) | Active Comparator (N=15)
Rehospitalization (Cardiac disorders) | 7 (15) | 7 (11)
Rehospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Rehospitalization (General disorders) | 1 (1) | 2 (2)
Rehospitalization (Renal and urinary disorders) | 0 (0) | 1 (1)
Rehospitalization (Surgical and medical procedures) | 0 (0) | 1 (1)
Rehospitalization (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rehospitalization (Nervous system disorders) | 0 (0) | 1 (1)
Rehospitalization (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Intervention (N=12) | Active Comparator (N=15)
ED visit (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ED visit (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ED visit (General disorders) | 2 (2) | 2 (3)
Urgent Care Visit (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes